CLINICAL TRIAL: NCT04167956
Title: Clinical Trial of Ultrasound Combined With Computed Tomography Guided Lumbar Sympathetic Ganglion Block for the Safety and Efficacy of Patients With Refractory Pain Caused by Sympathetic Neuropathy of Lower Extremities
Brief Title: Clinical Trial of Ultrasound Combined With Computed Tomography Guided Lumbar Sympathetic Ganglion Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: China-Japan Friendship Hospital (Other); First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ym20191016
Record Dates: First submitted 2019-10-17; First posted 2019-11-19 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-01

CONDITIONS: Pain, Chronic; Sympathetic Disorder; Ultrasound Therapy
Keywords: lumbar sympathetic; ultrasound
MeSH Terms: conditions — Chronic Pain; Autonomic Nervous System Diseases | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound combined with CT guided (Experimental): ultrasound combined with CT guided lumbar sympathetic ganglion block in patients with intractable pain caused by sympathetic neuropathy of lower extremities
  Interventions: Device: ultrasound and CT
- CT guided (Sham Comparator): CT guided lumbar sympathetic ganglion block in patients with intractable pain caused by sympathetic neuropathy of lower extremities
  Interventions: Device: ultrasound and CT

INTERVENTIONS:
Device: ultrasound and CT — Experimental: ultrasound combined with CT guided Active Comparator: CT guided

SUMMARY:
To evaluate the safety and efficacy of ultrasound combined with CT-guided sympathetic ganglion block for refractory pain caused by sympathetic neuropathy of the lower extremities.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of ultrasound combined with CT-guided sympathetic ganglion block for refractory pain caused by sympathetic neuropathy of the lower extremities. Patients with lumbar sympathetic block were enrolled and randomized to a conventional CT-guided group and an ultrasound-guided CT-guided group. By comparing the traditional CT guided and ultrasound combined with CT guided two programs, the radiation dose, block success rate, treatment time, etc. received by patients with lumbar sympathetic block were observed to understand whether ultrasound combined with CT guidance is a way to reduce radiation exposure. Under the premise of the dose, the method of blocking the success rate can still be guaranteed.

ELIGIBILITY:
Inclusion Criteria:

1.18~80 years old; 2.Pain disorders requiring lumbar sympathetic block（Such as,Lower limb vascular disfunction,Diabetic polyneuropathy,Postherpetic neuralgia,Complex regional pain syndrome I and II,Cancer related neuropathic pain including Peripheral neuropathy caused by chemotherapy or other lower extremity sympathetic neuropathy）,conservative treatment for 3 months or longer can not be cured; 3.Numerical rating score≥4.

Exclusion Criteria:

1. Body mass index> 30 kg / m2;
2. History of internal fixation in posterior lumbar laminectomy or any serious anatomic variation, such as scoliosis and tumors;
3. History of lumbar sympathetic neurochemistry or thermal neurolysis;
4. Pregnancy;
5. The puncture site is infected;
6. Coagulation dysfunction;
7. Allergic to local anesthetic or contrast agent;
8. Cognitive impairment or inability to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
The success rate of block | through study completion, an average of 7 days
  Numerical rating score（NRS） less than 4

SECONDARY OUTCOMES:
The skin temperature | 10 minutes
  The skin temperature
The toe perfusion index | 10 minutes
  The toe perfusion index
The number of patients satisfied with the first angiography | immediately
  The number of patients satisfied with the first angiography

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Doctor, Study Chair — Zhejiang University
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China